CLINICAL TRIAL: NCT06741709
Title: A Study of Mitral Annular Disjunction in Mitral Valve Prolapse Patients and Arrhythmia Risk
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Rezk Ayad Girgis, Resident doctor, Assiut University
Other Study IDs: Mitral annulus disjunction
Record Dates: First submitted 2024-10-24; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Mitral Valve Prolapse; Mitral Valve Insufficiency
Keywords: Mitral annular disjunction
MeSH Terms: conditions — Mitral Valve Prolapse; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the characteristics and prevalence of mitral annular disjunction in patients with mitral valve prolapse with severe mitral regurgitation (MR) at Assiut University Heart Hospital.

DETAILED DESCRIPTION:
Mitral annular disjunction is a structural defect of the mitral annulus fibrous commonly associated with mitral leaflet prolapse. However, there have been few cases of mitral annular disjunction in mitral valve prolapse (MVP).

Mitral annular disjunction (MAD) is a structural defect characterized by a clear separation between the mitral valve annulus, the left atrium wall, and the myocardial continuity. This condition can be seen in a 360-degree circle around the mitral valve annulus. However, it is most typically seen in the inferolateral myocardium, right behind the posterior mitral valve leaflet. It is generally present in the P1 and P2 mitral valve scallops.

Mitral valve prolapse (MVP) occurs in 3% of the population and is the most common reason for mitral valve replacement[1]. According to population and cohort studies, the patient's age significantly influences mitral valve prolapse (MVP) outcomes, left ventricular ejection fraction, and the severity of mitral regurgitation. Mitral regurgitation has little influence if it is not severe. While the link between MVP and sudden cardiac death was first discovered many years ago, it was once assumed to be extremely low risk. Recent observational studies have found a link between MVP and malignant ventricular arrhythmias, as well as sudden cardiac death, in a particular population of young and middle-aged people. This raise worries regarding the existence of an arrhythmic MVP variation. Recent research has led to a better knowledge of the aberrant physiological processes and circumstances that enhance the likelihood of developing irregular heart rhythms in people with mitral valve prolapse.

The diagnosis of mitral valve regurgitation can be accurately determined by non-invasive imaging techniques such as transthoracic echocardiography, Transesophageal echocardiography, and cardiac magnetic resonance imaging.

This study tries to improve patient risk assessment

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients > 18 years of age presenting to Assiut University Heart Hospital with MVP and more than moderate MR.

Exclusion Criteria:

* Previous mitral valve surgery.

  * MVP due to infective endocarditis.
  * Moderate or more significant aortic stenosis, aortic regurgitation or mitral stenosis.
  * Congenital heart disease and poor image quality precluding accurate assessment of the mitral valve.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-14 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Detect the prevalence of mitral annular disjunction in patients with mitral valve prolapse | six months
  Detect the prevalence of mitral annular disjunction in patients with mitral valve prolapse

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hussain N, Bhagia G, Doyle M, Rayarao G, Williams RB, Biederman RWW. Mitral annular disjunction; how accurate are we? A cardiovascular MRI study defining risk. Int J Cardiol Heart Vasc. 2023 Nov 9;49:101298. doi: 10.1016/j.ijcha.2023.101298. eCollection 2023 Dec. PMID 38035256
- [Background] Tison GH, Abreau S, Barrios J, Lim LJ, Yang M, Crudo V, Shah DJ, Nguyen T, Hu G, Dixit S, Nah G, Arya F, Bibby D, Lee Y, Delling FN. Identifying Mitral Valve Prolapse at Risk for Arrhythmias and Fibrosis From Electrocardiograms Using Deep Learning. JACC Adv. 2023 Aug;2(6):100446. doi: 10.1016/j.jacadv.2023.100446. Epub 2023 Aug 5. PMID 37936601
- [Background] Donal E, Galli E, Letourneau T. Need for expertise in mitral valve regurgitation. Open Heart. 2019 Apr 28;6(1):e001039. doi: 10.1136/openhrt-2019-001039. eCollection 2019. No abstract available. PMID 31168391
- [Background] Zoghbi WA, Adams D, Bonow RO, Enriquez-Sarano M, Foster E, Grayburn PA, Hahn RT, Han Y, Hung J, Lang RM, Little SH, Shah DJ, Shernan S, Thavendiranathan P, Thomas JD, Weissman NJ. Recommendations for Noninvasive Evaluation of Native Valvular Regurgitation: A Report from the American Society of Echocardiography Developed in Collaboration with the Society for Cardiovascular Magnetic Resonance. J Am Soc Echocardiogr. 2017 Apr;30(4):303-371. doi: 10.1016/j.echo.2017.01.007. Epub 2017 Mar 14. No abstract available. PMID 28314623